CLINICAL TRIAL: NCT01953614
Title: Effects of Chiropractic Adjustments on Brain Function Using Quantitative Encephalography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: I-0010
Record Dates: First submitted 2013-08-23; First posted 2013-10-01 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Brain Function
Keywords: quantitative encephalography; brain computer interface; chiropractic; sacro-occipital technique
MeSH Terms: interventions — Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Placebo group (Sham Comparator): Ten people. Participants will receive what appears to be a chiropractic adjustment but which actually is not. This is the sham adjustment. Participants will also fill out Achenbach questionnaire. There will be a follow up in 7 days.
  Interventions: Other: Sham adjustment
- Chiropractic adjustment (Active Comparator): Ten people. Group will be getting chiropractic adjustments. Participants will be filling out Achenbach questionnaire. There will be a follow up in 7 days.
  Interventions: Other: Chiropractic adjustment
- Control group (No Intervention): Ten people. This group will simply have their EEG recorded at baseline and after 7 days. There will be an Achenbach questionnaire like the two other groups.

INTERVENTIONS:
Other: Chiropractic adjustment
  Arms: Chiropractic adjustment
Other: Sham adjustment
  Arms: Placebo group

SUMMARY:
Despite the abundance of theories concerning the effects of chiropractic adjustments on brain function, this remains an understudies area for the profession.

Quantitative Electroencephalography (qEEG)is a technique that allows for an in-depth analysis of brain function. A normative database will be used to compare before, during and after effects of chiropractic adjustments on brain function. This will include usage of Low Resolution Electromagnetic Tomography (LORETA).

This study seeks to objectively document effects of chiropractic adjustments on brain function.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to receive chiropractic adjustments

Exclusion Criteria:

* No benzodiazepine class drugs in study participants
* No use of medicines such as Sudafed (pseudoephedrine) or Nyquil (Doxylamine succinate)
* At least 30 days since last chiropractic adjustment

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in quantitative EEG values as compared to a normative database | Baseline, during adjustment, after adjustment, follow up in 7 days
  There will be a baseline measurement. There will be measurements during the adjustment. There will be measurements immediately after the adjustment. There will be measurements 7 days after the adjustment.
  Data will then be analyzed comparing values to a normative database. This database is adjusted for age. This will generate z-score values in addition to raw EEG values. Statistical analysis of P-values will then be run to test significance of changes.

SECONDARY OUTCOMES:
Behavioral assessment questionaire | At baseline, one week after adjustment.
  Subject will be asked to complete the Achenbach System of Empirically Based Assessment. This assessment asks questions about subjects adaptive and maladaptive functioning. This information is comparing the subject to other people their age.

CONTACTS AND LOCATIONS:
Locations (1):
- Life University, Marietta, Georgia, United States